CLINICAL TRIAL: NCT06427551
Title: Peng Block in Total Hip Replacement: Effects of Anesthetic Volume on Clinical Outcome and Postoperative Complications
Brief Title: Volume Effect in Peng Block for Total Hip Replacement
Acronym: volupeng
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Serena Ricalzone, principal investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: VOLUPENG
Record Dates: First submitted 2024-04-26; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Post Operative Pain
Keywords: postoperative; orthopedic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 15 ml local anesthetic: in this group of patients the peng block was performed with 15 ml of ropivacaine, whose dose was obtained on the weight
  Interventions: Drug: Ropivacaine
- 20 ml local anesthetic: in this group of patients the peng block was performed with 20 ml of ropivacaine, whose dose was obtained on the weight
  Interventions: Drug: Ropivacaine
- 30 ml local anesthetic: in this group of patients the peng block was performed with 30 ml of ropivacaine, whose dose was obtained on the weight
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — The local anesthetic was dosed on the patient's weight (50-59kg: 120mg, 60-61kg: 140mg, 70-79kg: 160mg, ≥80kg: 180mg)

SUMMARY:
This study is to investigate whether a different volume of ropivacaine, with the same prescribed dosage based on body weight, can affect block efficacy, duration and side effects in the first 24 hours postoperatively.

DETAILED DESCRIPTION:
patients were divided into 3 groups on the basis of the volume of anesthetic given to perform the block. in every patient was assessed the nrs, the side effects, if any, and the need for analgesic drugs in the first 24 hour after surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA I, ASA II, ASA III
* Age≥18
* Total hip replacement surgery in spinal anesthesia
* Informed consent

Exclusion Criteria:

* ASA IV
* INR>1.3
* platelet values<100*10^3/ml a
* patients on anticoagulant or antiplatelet therapy
* general anesthesia for total hip replacement surgery
* patients on chronic opioid therapy
* altered sensitivity or motility
* Patients in chronic opioid therapy
* Refuse to sign informed consent form
* Unable to sign informed consent form
* Know allergies to medication used for analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent total hip replacement in elective surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
NRS evaluation | 24h post-op
  Evaluate pain for every volume group in the first 24 hours post surgery using the Numeric Pain Scale (NRS) assigning a numeric value between zero (no pain) and ten (the worst pain ever felt). Absence of relevant pain is considered a NRS less than three.
  Success of the block was defined as NRS≤3.

SECONDARY OUTCOMES:
NRS variation in time | 24 h
  consider variation of pain, assessed with numeric Pain scale, for each group, every six hours

OTHER OUTCOMES:
presence of side effects | 24 hours
  Monitoring the onset of side effects (nausea/vomiting/hypotension/dizziness/sensitive impareiment) in every group of patients in the first 24 hours every six hours
analgesic requirements | 24 hours
  requirement of analgesic to control the pain, assessed every six hours

CONTACTS AND LOCATIONS:
Overall Officials: manuela nicastro, MD, Study Director — aoupisa
Locations (1):
- Edificio 3 - Azienda Ospedaliero Universitaria Pisana Cisanello, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No